CLINICAL TRIAL: NCT01542424
Title: A Prospective, Multicentre, Open Label, Non-controlled, Observational, 24-week Study in Patients Using NovoMix® 30 (Biphasic Insulin Aspart 30) or Levemir® (Insulin Detemir) for Treatment of Type 1 or Type 2 Diabetes Mellitus in Macedonia
Brief Title: An Observational Study in Patients Using NovoMix® 30 or Levemir® for Treatment of Type 1 or Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-1763
Record Dates: First submitted 2012-02-24; First posted 2012-03-02 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- BIAsp 30 users
  Interventions: Drug: biphasic insulin aspart 30
- IDet users
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Prescribed at the discretion of the physician
  Groups: BIAsp 30 users
Drug: insulin detemir — Prescribed at the discretion of the physician
  Groups: IDet users

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate efficacy and safety of NovoMix® 30 (biphasic insulin aspart 30) or Levemir® (insulin detemir) in subjects with type 1 or 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Macedonian people with diabetes mellitus (Type 1 or Type 2)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Macedonian people with diabetes mellitus (Type 1 or Type 2)
Sampling Method: Non-Probability Sample
Enrollment: 1889 (Actual)
Dates: Start 2006-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
HbA1c (glycosylated haemoglobin)

SECONDARY OUTCOMES:
Percentage of subjects reaching HbA1c target of maximum 7.0%
Postprandial plasma glucose (PPG)
Fasting plasma glucose (FPG)
Change in body weight
Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Skopje, North Macedonia

REFERENCES:
- [Result] Dimitrovski, Cedomir and Smokovski, Ivica and Makrevska, Snezana and Mileva, Iskira and Kostojcinoska, Mira (2009) Significant Improvements in Glycaemic Control without Weight Gain with Insulin Detemir in Clinical Reality: Experience from Macedonian Clinical Practice. In: ADA Congress 2009, 05-09 June 2009, New Orleans, USA.
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com